CLINICAL TRIAL: NCT04606368
Title: Evaluation of the Safety and Efficacy of Sequential Use of Monopolar Radiofrequency Treatment on Lower Face and Submental Area for Fat Reduction and Improvement of Skin Laxity
Brief Title: Bausch Health Thermage FXL for Use on Lower Face and Submentum Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lorraine Hickson (Other)
Collaborators: Bausch Health Americas, Inc. (Industry); Solta Medical (Industry)
Responsible Party: Sponsor-Investigator, Lorraine Hickson, Director, Riverchase Dermatology
Organization: Riverchase Dermatology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bausch Health 2019-4816
Record Dates: First submitted 2020-10-12; First posted 2020-10-28 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Skin Wrinkling

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, non-randomized, interventional cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Interventional cohort (Experimental): Each subject will serve as their own control. Left side of lower jaw and submental area is control side. Right side of subject's lower jaw and submentum area will receive treatment.
  Interventions: Device: Thermage FLX

INTERVENTIONS:
Device: Thermage FLX — Monopolar radiofrequency will be applied through the Thermage FLX machine to the subject's right lower jaw and submentum area.

SUMMARY:
This study is designed to evaluate the safety and efficacy of sequential use of monopolar radiofrequency on lower face and submental area, followed by cryolipolysis on the submentum and submandibular area for fat reduction and improvement of skin laxity.

DETAILED DESCRIPTION:
This research study will study subjects who have mild to moderate skin laxity on lower jaw and submentum areas. This will be measured by conducting a treatment using the Thermage FLX system on the lower face and submentum area of the participants. Biopsies will be done on several locations throughout the 12 week trial to assess skin laxity through laboratory measures. Finally, the subject will be asked to complete questionnaires to provide satisfaction and tolerability feedback.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects > 40 years of age and < 80 years of age.
* Presence of mild to moderate skin laxity on lower face and submentum area, which in the investigator's opinion may benefit from monopolar radiofrequency to improve the skin laxity for a youthful, rejuvenated appearance.
* BMI under 35.
* Agreement to maintain their weight within 5 lb of the baseline.
* Subject has read and signed a written informed consent form.

Exclusion Criteria:

* Subject has severe skin laxity in the area of intended treatment which in the opinion of the investigator, may result in an unacceptable aesthetic result.
* Subject has had a surgical procedure(s) in the area of intended treatment.
* History of a fat reduction procedure (e.g., liposuction, surgery, lipolytic agents, etc.), in or around the area of intended treatment.
* Subject needs to administer, or has a known history of subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
* Currently taking or has taken diet pills or weight control supplements within the past month.
* Any dermatological conditions, such as scars, infection, in the location of the treatment area that may interfere with the treatment or evaluation.
* Active implanted device such as a pacemaker, defibrillator, or drug delivery system.
* Pregnant or intending to become pregnant in the next 6 months.
* Lactating or has been lactating in the past 6 months.
* BMI ≥ 35.
* Unable or unwilling to comply with the study requirements.
* Currently enrolled in a clinical study of any other unapproved investigational drug or device.
* Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-04-02 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent Adverse Events [Safety and Tolerability] | 12 weeks
  The primary objective of this study is to evaluate the safety and efficacy of improvement of skin laxity with the use of monopolar radiofrequency (Thermage FLX, Solta Medical) on lower face and submentum areas. Safety is defined as incidence of device- and/or procedure-related adverse events. Qualitative measurement of efficacy by independent blinded evaluators grading randomized baseline and 3 months follow-up photographs using a 4-point skin laxity rating scale.

SECONDARY OUTCOMES:
Subjective clinical evaluation of skin laxity with the use of monopolar radiofrequency treatment on lower face and neck [Efficacy] | up to 12 weeks
  Quantitative measurement of efficacy by standardized 2-D and 3-D images with volume difference in cc, height difference in mm, and surface area reduction measures calculations in cm2 using VECTRA H2 (Canfield Scientific, Inc), as well as, by histochemistry evaluation of punch biopsies performed at baseline, 4 weeks and 12 weeks post-procedure.
Subject satisfaction of skin laxity treatment on lower face and submentum areas documented in written questionnaire | though study completion, up to 12 weeks
  Subject satisfaction data will be collected at the 12-week final follow-up visit via a written questionnaire. A validated questionnaire using a likert rating scale will be utilized . Score values are 1 to 5, with high numbers meaning better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Leyda R Bowes, MD, Principal Investigator — Riverchase Dermatology
Locations (1):
- Riverchase Dermatology, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No